CLINICAL TRIAL: NCT00628459
Title: Effect of Iron Versus Multiple Micronutrient Supplementation on Anemia in Preschool Children of Malaria-Endemic Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre National de la Recherche Scientifique et Technologique (Other Government)
Collaborators: Université Libre de Bruxelles (Other); Fonds pour la recherche scientifique médicale (FRSM), Belgium (Unknown)
Responsible Party: Hermann Ouédraogo, chargé de recherche, Institute of Research in Health Sciences
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MIENKO2
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Last update posted 2008-03-05 (Estimated); Status verified 2008-02

CONDITIONS: Anemia; Undernutrition
Keywords: iron; multiple micronutrient; malaria; anemia; preschool children
MeSH Terms: conditions — Anemia; Malnutrition; Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator)
  Interventions: Dietary Supplement: micronutrient supplementation
- 2 (Experimental)
  Interventions: Dietary Supplement: micronutrient supplementation
- 3 (Experimental)
  Interventions: Dietary Supplement: micronutrient supplementation

INTERVENTIONS:
Dietary Supplement: micronutrient supplementation — Supplements are given daily, 5days/week, for 6 months, involving 15 mg iron (arm 1), 15 mg iron and 10 mg zinc (arm 2), or multiple micronutrient (arm 3): 15 mg iron, 10 mg zinc, 375 µg vitamin A, 5 µg vitamin D, 6 mg vitamin E, 0.5 mg vitamin B1, 0.5 mg vitamin B2, 6 mg niacin, 150 µg folic acid, 0.5 mg vitamin B6, 0.9 mg vitamin B12, 35 mg vitamin C, 10 µg vitamin K, 50 µg iodine, 0.6 mg copper.

SUMMARY:
Some micronutrients are likely to interact with malaria parasite, leading to either synergistic or antagonist effect on malaria morbidity and therefore on hemoglobin response.

The purpose of this study is to investigate the effect of supplementation with iron or multiple micronutrients on anemia while integrated with malaria management in rural Burkinabe young anemic children with high prevalence of malaria.

DETAILED DESCRIPTION:
This is a community-based randomised double-blind trial. Children aged 6-23 months are randomised to receive either iron (n=91), iron and zinc (IZ, n=90) or MMN (n=89), 5 days/week for 6 months. Supplements are manufactured by Nutriset (Malaunay, France) as specifically fortified "plumpy-nut". They are presented in 90 ml boxes coded A, B and C each lot of boxes contained in white packing labelled A, B and C respectively. Malaria is managed in concordance with the national malaria program standards. All mothers receive one insecticide-treated bed-net (PermaNet®, Vestergaard Frandsen Disease Control Textiles) and instruction for effective utilization for children. All children with positive smear for Plasmodium falciparum are artemether+lumefantrine-treated (Coartem®, Novartis Pharma S.A.S., France) regardless of the clinical status. Children aged of at least 12 months receive 200 mg albendazole, one week prior to the supplementation starting.

Data collection involves:

* a questionnaire addressed to mothers at baseline,
* a medical examination of mothers and children at baseline: A general practitioner examines mothers for goiter determination according to the International Council for the Control of Iodine Deficiency Disorders (ICCIDD) definition and classification, and children for splenomegaly that is classified according to Hackett. Anthropometrical measurements are performed on children and mothers by a nutritionist, in agreement with the WHO recommendations. Children's capillary blood is obtained by lab technicians through a finger stick for hemoglobin measurement and malaria blood smear preparation. Hemoglobin is measured using a HemoCue® machine (Hemocue HB 201+, Angelholm, Sweden) to the nearest 1g/L.
* malaria microscopic detection at baseline and monthly during the study: blood smears intending to detect malaria infection are stained with Giemsa, and read in duplicate at the local hospital laboratory,
* a daily record of supplementation and morbidity data (diarrhoea, fever, cough).

The endpoints considered for analysis are change of hemoglobin (final haemoglobin minus baseline haemoglobin concentration) and final anemia status that are analysed by multiple linear regression and logistic regression respectively.

ELIGIBILITY:
Inclusion Criteria:

* age of 6-23 months
* hemoglobin concentration range of 70-109 g/L

Exclusion Criteria:

* severe wasting (weight-for-height z-score < -3)

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 297 (Actual)
Dates: Start 2006-08; Primary Completion 2007-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Anemia | 6 months

SECONDARY OUTCOMES:
Growth | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Donnen, PhD, Study Director — Université Libre de Bruxelles, Belgium
Locations (1):
- District Sanitaire de Kongoussi, Kongoussi, Burkina Faso

REFERENCES:
- [Background] Smuts CM, Dhansay MA, Faber M, van Stuijvenberg ME, Swanevelder S, Gross R, Benade AJ. Efficacy of multiple micronutrient supplementation for improving anemia, micronutrient status, and growth in South African infants. J Nutr. 2005 Mar;135(3):653S-659S. doi: 10.1093/jn/135.3.653S. PMID 15735110